CLINICAL TRIAL: NCT01911208
Title: A Randomized Recruitment Intervention Trial
Acronym: RECRUIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Barbara Tilley, SPH Faculty - Biostatistics, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIMHD006941; U24MD006941 (NIH)
Record Dates: First submitted 2013-01-24; First posted 2013-07-30 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Recruitment of Minorities
Keywords: Minority; Recruitment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RECRUIT intervention (Experimental): Clinical sites will work with the RECRUIT team to enhance and individualize their recruitment methods.
  Interventions: Behavioral: RECRUIT intervention
- Control (Experimental): Clinical sites can use which ever recruitment methods they prefer.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: RECRUIT intervention — Sites randomized to RECRUIT are taught skills to develop a tailored recruitment intervention encompassing continuous quality improvement and patient navigation.
  Arms: RECRUIT intervention
Behavioral: Control — Non-intervention control.
  Arms: Control

SUMMARY:
The purpose of this study is to test a recruitment intervention to increase racial and ethnic diversity in clinical trials. The trial will be conducted in specialty care clinics. In RECRUIT minorities are those underrepresented in clinical trials and include:

* African Americans/ Blacks
* Asians
* Native Hawaiians/Other Pacific Islanders
* Hispanic/Latinos
* Native Americans/Alaskan Natives

DETAILED DESCRIPTION:
Low minority participation in clinical trials limits our ability to assess and address potential differences in therapeutic responses. To address the problem of low minority recruitment we are initiating a randomized trial of a recruitment intervention (RECRUIT) funded by the National Institute on Minority Health and Health disparities (NIMHD) to increase racial/ethnic diversity in clinical trials.

Our specific approach is directed toward multi-site trials conducted at specialty clinics within academic centers with recruiting venues that include community practices or practices of colleagues in other areas of the academic center. The intervention will focus on approximately 60 specialty clinics. Clinical sites will be randomized to the intervention or control group. The target of the intervention will be the site investigators and clinical trial coordinators.

ELIGIBILITY:
Inclusion:

A parent trial must :

* have a coordinating Center willing to allow their Clinical Sites to participate;
* be studying be studying a condition that requires community or health system physician referral
* be studying an intervention where the recruitment approach cannot be made directly to minority community members
* need to increase recruitment of racially/ethnically diverse participants* to the trial as demonstrated by current trial progress or historical data from other trials in the same disease;
* be a Phase II or Phase III trial
* be conducted in at least six multiple sites;
* expect each Clinical Site to recruit at least 10 participants;
* be funded by a sponsor (NIH or pharmaceutical company or other) that has a strong commitment to recruiting racially/ethnically diverse subjects;
* be willing to have investigators and coordinators attend a special training meeting (at RECRUIT expense);
* require randomization to intervention or control (could be best medical care or active control or placebo or other type of control);
* provide transportation costs for trial participants who need assistance in getting to trial sites or use some RECRUIT reimbursement for this purpose.

The clinical site must

* be a funded Clinical Site in the parent trial;
* be located in an area where at least 20% of the population within 30 miles in the age group under study in the parent trial are from diverse populations.

Exclusion Criteria:

* site does not agree to be randomized;
* investigator or coordinator is under 18 years of age.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
Percentage of racially/ethnically diverse participants (minorities) enrolled | Up to 2 years
  Minorities as defined in this trial include those underrepresented in clinical trials and considered underrepresented by NIH criteria with the addition of those of Asian descent.

SECONDARY OUTCOMES:
Number of participant referrals | up to 2 years
  Differences between intervention and control sites in number of participant referrals.
Recruitment Activities | up to 2 years
  Numbers and types of activities reported on recruitment logs by all sites.
Investigator and Coordinator Outcome expectations | up to 2 years
  Change from baseline in physician investigator and coordinator outcome expectations (intervention sites only).
Qualitative Key Informant Interviews | up to 2 years
  Qualitative key informant phone interviews of the physician investigators and coordinators (intervention and control sites).
Participant Satisfaction | up to 2 years
  Potential/enrolled participant satisfaction with intervention and control trial site investigators and coordinators. Subjects will be given a satisfaction survey at screening and at every follow up visit.
Investigator and Coordinator Self-Efficacy | up to 2 years
  Change from baseline in physician investigator and coordinator self-efficacy(intervention sites only).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara C. Tilley, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center School of Public Health, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tilley BC, Mainous AG 3rd, Amorrortu RP, McKee MD, Smith DW, Li R, DeSantis SM, Vernon SW, Koch G, Ford ME, Diaz V, Alvidrez J; additional RECRUIT Trial Center and Parent Trials' investigators. Using increased trust in medical researchers to increase minority recruitment: The RECRUIT cluster randomized clinical trial. Contemp Clin Trials. 2021 Oct;109:106519. doi: 10.1016/j.cct.2021.106519. Epub 2021 Jul 30. PMID 34333138
- [Derived] DeSantis SM, Li R, Zhang Y, Wang X, Vernon SW, Tilley BC, Koch G. Intent-to-treat analysis of cluster randomized trials when clusters report unidentifiable outcome proportions. Clin Trials. 2020 Dec;17(6):627-636. doi: 10.1177/1740774520936668. Epub 2020 Aug 24. PMID 32838555